CLINICAL TRIAL: NCT00217867
Title: A RCT to Reduce Cardiopulmonary Rehospitalization
Brief Title: Educational and Supportive Interventions to Prevent Cardiopulmonary Rehospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Brian Jack, faculty member, BMC, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-25057; R01HL081307 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (No Intervention): Usual Care, defined as the usual hospital discharge process as delivered by nurses and doctors.
- 2 (Experimental): Use of animated computerized character to prepare subjects for discharge by reviewing information provided to subjects in a printed After Hospital Care Plan packet, followed by telephone system to reinforce the discharge.
  Interventions: Behavioral: Animated character intervention with telephone follow-up

INTERVENTIONS:
Behavioral: Animated character intervention with telephone follow-up — Animated character will teach the discharge plan before discharge, then this teaching will be reinforced by computerized telephone system.
  Arms: 2

SUMMARY:
This study will use a comprehensive hospital discharge toolkit to implement up-to-date guidelines for cardiopulmonary diseases. The study will also include a computer-based patient-education program and a telephone-based post-discharge program, both designed for individuals with limited health literacy. The purpose of this study is to reduce early hospital readmission.

DETAILED DESCRIPTION:
BACKGROUND:

Limited health literacy is prevalent in America and has been identified as a cross-cutting priority area for transforming health care quality. This study will explore the effect of innovative patient-education and self-management systems on early rehospitalization for patients admitted to a general medical service.

DESIGN NARRATIVE:

This is a two-armed randomized study of patients with chronic cardiopulmonary diseases in three levels of health literacy. Patients will be tested with the 66 word version of the Rapid Estimate of Adult Literacy in Medicine (REALM) test to allow us to analyze the data according to literacy categories ( 6th grade, 7th-8th grade, and 9th grade). Patients will be randomized to one of the following groups: 1) standard discharge (control group); 2) a experimental group receiving both the case management intervention plus educational and self-management support by Embodied Conversational Agents (ECAs) and post-discharge reinforcement of the discharge plan using a computerized telephone system

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the general medical service at Boston Medical Center (BMC)
* Desires to be hospitalized in the future if there is a clinical need
* Able to communicate in English with health providers

Exclusion Criteria:

* Transferred from an outside hospital or a specialty services at BMC (e.g., orthopedic surgery, obstetrics and gynecology, otolaryngology, general surgery, or psychiatry)
* Requires hospice, nursing home, or other institutional settings
* Vision that is inadequate to discern the computer-based education and self-management support system
* Hearing that is inadequate to use a telephone
* Unable to independently consent
* Scheduled admission (e.g. for surgery)
* Has sickle cell disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 832 (Actual)
Dates: Start 2008-10; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Rehospitalization | Measured at 30 days

SECONDARY OUTCOMES:
Subject satisfaction with intervention and hospital experience | Measured at discharge and 30 days
Subject readiness for discharge | Measured at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Brian Jack, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States